CLINICAL TRIAL: NCT05954754
Title: The Effect of Diaphragmatic Breathing Exercises on Fetal Anxiety and Coping With Prenatal Stres
Brief Title: The Effect of Diaphragmatic Breathing Exercises on Fetal Anxiety and Coping With Prenatal Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sümeyye Barut, Assitant Professor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/3797
Record Dates: First submitted 2023-07-06; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Coping With Prenatal Stress; Fetal Health Anxiety
Keywords: Pregnancy,; breathing exercises,; fetal anxiety,; stress,; coping

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial
Who Masked: Participant
Masking Description: This study was designed as a randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic breathing exercise (Experimental): Diaphragmatic breathing exercise training was given individually to each pregnant women in the experimental group by one of the trained researchers. Two weeks after the first application, the researcher made the pregnant woman repeat the application 2 days a week via video call. Thus, a total of five diaphragmatic breathing exercises were applied to pregnant women in the experimental group during two weeks. They continued to do breathing exercises for 20-30 minutes a day for ten minutes each day for two weeks as they could tolerate.
  Interventions: Other: Diaphragmatic Breathing Exercises
- Control (No Intervention): The researchers applied no initiative to the control group, and the women in the control group solely had the routine checks. The women in the control group filled out all pretest forms(Personal Information Form,Revised-Prenatal Coping Inventory (NuPCI), Fetal Health Anxiety Inventory (FHAI)) were re-administered 2 weeks later to women who did not receive any intervention.

INTERVENTIONS:
Other: Diaphragmatic Breathing Exercises — Diaphragmatic breathing exercise training was given individually to each pregnant women in the experimental group by one of the trained researchers. Two weeks after the first application, the researcher made the pregnant woman repeat the application 2 days a week via video call. Thus, a total of five diaphragmatic breathing exercises were applied to pregnant women in the experimental group during two weeks. They continued to do breathing exercises for 20-30 minutes a day for ten minutes each day for two weeks as they could tolerate.
  Arms: Diaphragmatic breathing exercise

SUMMARY:
Objective: This study was conducted to determine the effect of diaphragmatic breathing exercises on coping with fetal anxiety and prenatal stress during pregnancy.

Methods: This randomized controlled study was carried out at a family health center in eastern Turkey. The study sample consisted of 106 pregnant women (experimental group, 54; control group, 54). Those in the experimental group received diaphragmatic breathing exercises five times in two weeks, one time via face-to-face session and 4 times twice a week via video call. Those in the control group received no intervention. Data were collected using the Revised-Prenatal Coping Inventory (NuPCI) and the Fetal Health Anxiety Inventory (FHAI).

DETAILED DESCRIPTION:
Introduction Pregnancy is a natural event that many women look forward to have with happiness and excitement, but it can be challenging for some women. In addition to physiological and psychological changes occurring during pregnancy, the readiness for a new life, changes in body image perception, fear of becoming a parent, uncertainties about childbirth, fears about the baby's development and survival can cause stress in pregnant women. Moreover, stressors during pregnancy such as economic problems, epidemics, and natural disasters can contribute to anxiety about both maternal and fetal health and cause significant stress. Stress is commonly observed during pregnancy and ranks high among stressful life events.

The negative effects of stress on human health are well-known. Both maternal and fetal health and their immune responses are sensitive to stress during pregnancy. High cortisol levels can lead to changes in their immune responses, suppressing the immune system and causing complications such as premature birth. Stress during pregnancy has been associated with negative pregnancy outcomes such as spontaneous abortion, pregnancy-induced hypertension, placental abnormalities, difficult labor, operative deliveries, low APGAR score, low birth weight, fetal death, postpartum depression, and long-term health problems such as cerebral palsy, neurodevelopmental delay, vision and hearing problems.

Although many pregnant women are exposed to stress, not all women who experience stress have negative pregnancy outcomes. The positive or negative experiences of pregnant women during pregnancy, their styles of coping with these experiences and stress, and the stressors they are exposed to affect whether the stress will disrupt their body balance and cause negative outcomes such as illness. The style of coping with stress is determinant in adapting to stressful events. Functional styles of coping with stress can reduce negative effects of stress, while ineffective coping styles can increase health risks. Coping styles of pregnant women with stress may vary, including functional coping styles such as having self-confidence, seeking social support, planning, and spiritual readiness and ineffective coping styles such as helplessness and avoidance. Considering the importance of coping with stress, understanding how pregnant women cope with stress and intervening to develop their styles of coping with stress may be useful in reducing stress during pregnancy. Various non-pharmacological methods such as relaxation exercises, yoga, biofeedback, massage therapy, acupuncture, and music therapy may be useful in reducing stress during pregnancy. However, there is no study about the effect of non-pharmacological methods in pregnancy on coping styles with stress. Some studies have reported that diaphragmatic breathing exercises increase quality of life and oxygenation and have a positive effect on anxiety. Therefore, both physical and psychological effects of diaphragmatic breathing exercises in pregnant women may positively affect their styles of coping with stress and reduce fetal anxiety. For this reason, this study aimed to determine the effect of non-pharmacological methods, specifically diaphragmatic breathing exercises, on coping with fetal anxiety and prenatal stress.

Research Hypothesis:

H1. Diaphragmatic breathing exercises performed during pregnancy increase coping with stress and reduce fetal health anxiety.

Method Design This randomized controlled study was conducted with pregnant women who were randomly assigned to experimental and control groups, and those who were assigned to the experimental group received diaphragmatic breathing exercises.

Sample The sample for the study consisted of pregnant women who referred to a family health center (FHC) in the center of a city in eastern Turkey. Healthy pregnant women were monitored by midwives and family physicians at the FHC, while high-risk pregnancies were referred to hospitals. There were no breathing exercise programs for pregnant women at the center.

The inclusion criteria for this study were as follows: (1) being pregnant women in their second and third trimesters (between 28-36 weeks); (2) being ≥18 years old; (3) having no medical pregnancy complications; (4) having no diagnosed mental illness; (5) having no fetal anomaly diagnosis; (6) using a smartphone.

A web-based software program was used to calculate the sample size for the study, considering the mean coping with stress during pregnancy score, which was the primary dependent variable. The coping with stress during pregnancy score reported by Faramarzi et al. was used as a reference (mean = 2.28, standard deviation = 0.54). The sample size was calculated to be 54 for each group (54 for the experimental group, 54 for the control group), assuming a 1-point increase in the mean coping with stress during pregnancy score after the intervention, with a two-sided significance level of 5%, 95% confidence interval, and 80% power. Randomization was used to assign pregnant women to either the intervention or control group. The Numbers section of the random.org website was used for randomization, and pregnant women who applied to the FHC were assigned to groups based on their order of arrival to the FHC, with the first and second women assigned to the experiment and control groups, respectively. The groups were allocated by a draw, where the number 1 was assigned to the experiment group and the number 2 was assigned to the control group. The same method was used to assign pregnant women to the experimental or control group until the desired sample size was reached.

Measures The data were collected by the researchers after routine check-ups of pregnant women between November 2022 and April 2023. After pregnant women were informed about the study, the researchers asked questions to those who agreed to participate in the study, and their answers were marked on the data collection forms. The primary outcome of the study, coping with stress during pregnancy, was evaluated using the Revised-Prenatal Coping Inventory (NuPCI). The secondary outcome, fetal anxiety, was measured using the Fetal Health Anxiety Inventory (FHAI).

A personal information form was created by the researchers in line with the literature to determine pregnant women's sociodemographic (age, education level, employment status, and income level) and pregnancy characteristics (trimester, gravida, and planned pregnancy).

The NuPCI was developed in 2020 and its Turkish validity and reliability study was conducted in 2022. The scale measures pregnant women's coping styles and perceptions of stress. It consists of 30 items and three subscales: Planning-preparation, Avoidance, and Spiritual-positive. This is a 5-point Likert-type scale, scoring from 0 (never) to 4 (very often). Higher planning-preparation and spiritual-positive subscale scores and lower avoidance subscale scores indicates higher coping with stress. Cronbach's alpha reliability coefficient for the planning-preparation, avoidance, and spiritual-positive subscales as 0.83, 0.57, and 0.69, respectively.

The FHAI was developed in 2019 and its Turkish validity and reliability study was conducted in 2022. The scale measures pregnant women's anxiety related to the fetus' health. It consists of 14 items, and each item consists of four statements that best capture the women's experiences in the previous weeks. This is 4-point Likert-type scale, scoring from 0 (no symptoms) to 3 (severe symptoms). The sum of item scores gives the total fetal health anxiety score, and as the total score increases, the level of fetal health anxiety also increases. The Cronbach's alpha reliability coefficient of the scale was 0.85.

Intervention In the present study, the pretest data were collected by the researchers through face-to-face interviews in the counseling room of the FHC. Two weeks later, the post-test data were obtained using the same method. After the pretest, diaphragmatic breathing exercise training was given individually to each pregnant women in the experimental group by one of the trained researchers, named E.S.B. At the end of the training, the pregnant women performed the exercise individually under the supervision of the researcher. Data collection, training and application lasted around 40 minutes. Two weeks after the first application, the researcher made the pregnant woman repeat the application 2 days a week via video call. The video calls were made on the day and time when pregnant women were suitable, and each application lasted around 10 minutes. Thus, a total of five diaphragmatic breathing exercises were applied to pregnant women in the experimental group during two weeks. They continued to do breathing exercises for 20-30 minutes a day for ten minutes each day for two weeks as they could tolerate. Although the optimal application time of breathing exercises is not yet determined in the literature, 2-3 sessions a week are planned for outpatients, while 5 sessions a week can be planned for inpatients. No intervention was applied to pregnant women in the control group by the researchers.

In order for pregnant women to apply the correct technique in diaphragmatic breathing exercises, they were asked to first rest for 1-2 minutes in a supine position with pillows under their heads and support from their knees on a flat surface. Their one hand was placed on the abdomen and the other on the upper part of the chest wall. While inhaling, their hand on the abdomen moved upwards, while the other hand remained as still as possible. While exhaling, their hand on the abdomen moved downwards, while the other hand remained as still as possible. They were asked to breathe quickly, deeply, and without causing fatigue. They were told to breathe through the nose and exhale through the mouth. To prevent the risk of hyperventilation, they were instructed to slowly exhale all the air using controlled expiration. After they performed diaphragmatic breathing exercises correctly, the exercises were repeated in a sitting position. In the two-week exercise program, the exercises were performed in a seated position.

Statistical analysis For the statistical analysis, the data were assessed using SPSS 25.0 for Windows software (SPSS, Chicago, IL, USA). Descriptive statistical values, numbers, percentages, means and standard deviations were used for the analysis. Comparisons of the categorical variables between groups were carried out using the chi-squared test. An independent-samples t-test was used to make comparisons between the experimental and control groups; a paired-samples t-test was used to make comparisons intra-groups. If the results of the t-tests were significant, effect sizes were computed using Cohen's d to identify significant differences. The statistical significance level was considered as p < 0.05.

Ethics For conducting the study, an ethical approval was obtained from the Fırat University Health Sciences Non-Invasive Clinical Research and Publication Ethics Committee (Decision No: 2022/3797). Pregnant women were informed about the purpose and method of the study, and a written informed consent form was obtained from those who agreed to participate in the study. After the data collection phase was completed, a single session breathing exercise training was given to the pregnant women in the control group for approximately 30-40 minutes.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant women in their second and third trimesters (between 28-36 weeks);
* being ≥18 years old;
* having no medical pregnancy complications;
* having no diagnosed mental illness;
* having no fetal anomaly diagnosis;
* using a smartphone.

Exclusion Criteria:

* Diagnosis of any chronic disease and initiation of medication for chronic disease during the research process
* Detection of fetal congenital malformation in the research process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — being ≥18 years old
Enrollment: 108 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Revised-Prenatal Coping Inventory (NuPCI) | Change from Revised-Prenatal Coping Inventory at 2 weeks
  The scale measures pregnant women's coping styles and perceptions of stress. It consists of 30 items and three subscales: Planning-preparation, Avoidance, and Spiritual-positive. This is a 5-point Likert-type scale, scoring from 0 (never) to 4 (very often). Higher planning-preparation and spiritual-positive subscale scores and lower avoidance subscale scores indicates higher coping with stress.

SECONDARY OUTCOMES:
Fetal Health Anxiety Inventory (FHAI) | Change from Fetal Health Anxiety Inventory at 2 weeks
  The scale measures pregnant women's anxiety related to the fetus' health. It consists of 14 items, and each item consists of four statements that best capture the women's experiences in the previous weeks. This is 4-point Likert-type scale, scoring from 0 (no symptoms) to 3 (severe symptoms). The sum of item scores gives the total fetal health anxiety score, and as the total score increases, the level of fetal health anxiety also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No